CLINICAL TRIAL: NCT04207476
Title: Effects on Autonomic Nervous System Through Utilization of an Electromagnetic Resonator in Heart Failure
Brief Title: Magnesphere for Autonomic Alteration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated due to COVID and computer difficulties.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11415
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment arm (Experimental): Active magnetic field exposure will be performed by use of a EMF resonator. Stimulator will be applied continuously for 1 hour.
  Interventions: Device: EMF
- Placebo (Placebo Comparator): Placebo magnetic field exposure will be performed by use of a EMF resonator. Stimulator will be applied continuously for 1 hour.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: EMF — Active magnetic field exposure will be performed by use of a EMF resonator. Stimulator will be applied continuously for 1 hour.
  Arms: Treatment arm
Device: Placebo — No magnetic field exposure will be given while patients are assigned to this arm for a duration of 1 hour.
  Arms: Placebo

SUMMARY:
To evaluate the physiologic effects of an electromagnetic resonator(EMF) on autonomic nervous system tone modulation through measurement of heart rate variability(HRV).

Null Hypothesis: An EMF Resonator will not change autonomic nervous system tone and no demonstrable difference in physiological parameters will recorded.

Alternative Hypothesis: Using an EMF Resonator will enhance parasympathetic activty as supported by HRV.

DETAILED DESCRIPTION:
During the initial encounter, participants will be randomized to either therapy or sham. The randomization scheme will be blinded to all investigators, will be devoid of patient information, and will be programmed by a non·investigator third party. All patients will receive the same total duration of therapy, and all patients will receive a sham and a treatment session.

Participants will wear head phones to reduce effects of any outside noises and will lay supine in a chair at approximately 40 degrees which is inside the FDA approved Resonator® EMF field. The active treatment session will be A160 which is a narrow range but variable magnetic field. This ranged from 3.1 x10·8 to 3.2 x 10-8 amplitude with a frequency of 0.857-0.859.

Eligible participants will arrive for testing in the morning and will be randomized to either treatment sequence. Randomization will be predetermined. Mobile phones and pagers will be placed into airplane mode during the study on a table in the room. The patient will be connected to HRV measurement systems. A BP reading will be taken in each arm. Patients will then lay supine in a standardized relaxation chair at approximately 40 degrees at which time the headphones will be placed. Ambient room light will remain powered on during therapy and will remain unchanged regardless of randomization. The researcher will then start either arm A or B (based on randomization). During the session, each participant will be given a short novel/magazine to read to reduce the chance of sleeping.

All HRV monitors will be disconnect and the subject's electronics will be returned.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients more than 18 years old with LVEF of < 40%(N=20)
2. Healthy age matched controls (N=20)
3. Ability to lay in a reclining chair for at least 60 minutes

Exclusion Criteria:

* 1. Inability to provide consent 2. Significant valvular disorder (i.e., prosthetic valve or hemodynamically relevant valvular diseases) 3. Recent (<6 months) stroke or myocardial infarction 4. Severe heart failure (NYHA IV) 5. Hemodialysis 6. Recurrent vaso-vagal syncopal episodes 7. Unilateral or bilateral vagotomy 8. Pregnancy or breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-25 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Heart rate variability(HRV) | 1 hour
  HRV will be measured using continuous 10 minute ECG pre and post exposure

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Dasari, MD, Principal Investigator — OUHSC
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No